CLINICAL TRIAL: NCT07205978
Title: Nut Consumption and Prevention of Non-communicable Diseases: A Global Individual Participant Data Meta-analysis
Acronym: NUTPOOL
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jordi Salas, Professor and Co-Prinicpal Investigator NUTPOOL, Institut Investigacio Sanitaria Pere Virgili
Other Study IDs: NUTPOOL
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetes (DM); Cardio Vascular Disease; Cancer; Dementia; Dementia Alzheimer Type; Mortality; Parkinson Disease (PD); Death
Keywords: nuts; moratlity; cardiovascular disease; Diabetes; dementia; IPD; epidemiology; Tree nuts; Peanuts; walnuts; almonds; pistachios; macadamia; cashewnut; pine nuts; Brazil nuts; Adult; Type-2 diabetes, Diabetes Mellitus, type 1*; Cardiovascular diseases*; Coronary health disesase; Alzheimer disease*; Parkinson disease*; Mortality*; Death*; Fatal outcome*; nut
MeSH Terms: conditions — Diabetes Mellitus; Neoplasms; Dementia; Alzheimer Disease; Parkinson Disease; Death; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The proposed aims will be evaluated using data from prospective cohort studies from around the world: Prospective studies will be eligible if they have good quality nutrition data from a food frequency questionnaire (FFQ) about total nuts and/or specific nuts, and well-ascertained data of at least two of the health outcomes (T2D, CVD, cancer, or dementia), more than 1,000 adult participants, and accrued five years or more of median follow-up that allows time-dependent analyses. We expect 25-30 cohorts to be included in the final analysis.

SUMMARY:
The relationship between nut consumption and the risk of developing non-communicable diseases (NCDs) has been a subject of growing interest. However, the findings from previous studies have been conflicting for some health outcomes, such as type-2 diabetes, and have been underexplored for other outcomes, such as neurodegenerative diseases. One contributing factor to these inconsistencies lies in the different analytical approaches and confounding factors used across studies. Furthermore, the majority of previous studies have primarily focused on populations in Europe or the United States, potentially limiting the generalizability of the findings to other global regions. The NUTPOOL project aims to address these gaps by conducting an extensive individual participant data (IPD) meta-analysis. This study will evaluate the association between total and specific types of nut consumption and the future risk of NCDs.

DETAILED DESCRIPTION:
NCDs account for 74% of global deaths, with 41% of these occurring prematurely in individuals aged 70 years and older. Type 2 diabetes, cardiovascular diseases (CVD), and cancer are among the major chronic diseases that affect people across countries and contribute to premature deaths. Notably, 77% of all NCD deaths and 86% of premature deaths occur in low- and middle-income countries. Reducing premature mortality from NCDs through preventive strategies, especially in low- and middle-income countries, was identified as a target in the Sustainable Development Goals from the World Health Organization. Additionally, as populations age, dementia is gaining recognition as a major public health concern. Dementia is among the leading causes of death and disability, with significant economic implications. Therefore, implementing preventive strategies to maintain cognitive function and delay cognitive decline is essential.

Adhering to a healthy diet is an effective and cost-efficient strategy to reduce NCDs. In fact, unhealthy diets have been linked to over 30% of NCDs and cognitive decline. Nuts are a common food component of several plant-based diets that have shown beneficial effects in preventing NCDs. Nuts are a diverse food group comprising a wide variety of oily kernels with a unique nutritional profile, including high amounts of protein, fiber, unsaturated fatty acids, vitamins, polyphenols, and other phytochemicals. These nutrients may contribute to their beneficial effects, such as antioxidant, anti-inflammatory, antihypertensive, anti-lipidemic, and anti-aging properties, as well as their potential positive influence on gut microbiota modulation.

Prior research has examined the impact of nuts on various health outcomes; however, many of these studies have focused on intermediate outcomes, obtained controversial results, and have been conducted primarily in European countries or the United States. Furthermore, the data has been analyzed using a variety of approaches, the studies were designed in different ways, and different covariates were added to the statistical models, potentially leading to inconsistencies and compromising the reliability of the comparison between studies. These inconsistencies emphasize the need for further research to elucidate the role of total nuts and specific types of nut consumption on the development of highly prevalent NCDs, as well as to allow the generalizability of the results across different countries and ethnicities.

In the NUTPOOL project, the objective is to address these knowledge gaps and provide a thorough assessment of the associations between total nuts and specific types of nuts in relation to a wide range of NCDs and mortality. The results from this global collaborative project will be representative of the worldwide populations, as they include prospective cohort studies from different countries, including not only American and European countries, but also Asian and Oceania. Additionally, the focus is on total and specific types of nuts, along with highly prevalent and relevant outcomes such as type 2 diabetes, cardiovascular disease (CVD), cancer, dementia, and mortality. To ensure consistency and reliability, the analyses will be standardized using Individual Participant Data (IPD) meta-analyses.

The selection of studies will be conducted after the identification of cohorts with data available on nut consumption. This identification process will be based on information comprehensively extracted from recently published systematic reviews and meta-analysis (SRMAs) on the subject, as well as through extensive research network. Invitations will be extended to as many eligible cohorts as possible to mitigate selection bias and ensure comprehensive participation in the study. Studies will be eligible for inclusion if they reported reliable nutrition data from a food frequency questionnaire (FFQ) regarding total nuts and/or specific nuts, along with well-defined data on at least two of the health outcomes. The study population had to be at least 1,000 adults, and the study had to span a minimum of five years or more of median follow-up, enabling time-dependent analyses.

The assessment of nut consumption involves standardizing the amount consumed to a standard serving size (1 serving = 28 g or 1 oz.). The cumulative average or baseline nut consumption will be used according to the data collection methods employed for each cohort. Nut consumption will be analyzed as both a continuous and a categorical variable. The methods used to ascertain high-prevalence NCDs include medical diagnosis, official national or regional death registers, self-reported cases, and medication checks.

The statistical analysis plan will entail the subsequent two steps: First, each cohort will follow a standardized and harmonized protocol to analyze the data. Secondly, centralized meta-analyses will be performed. Multivariable Cox proportional hazards models will be used to estimate the risk of NCDs. Separate models will be conducted for categories of total nuts and specific types of nuts. A dose-response analysis will also be conducted. The models will include different levels of adjustment:

* Model 1: age and sex
* Model 2: M1 + race, family history of NCDs of interest, personal history of hypercholesterolemia, education level, physical activity, alcohol consumption, smoking, total energy intake, cohort specific adjustements (e.g. allocation to intervention group for intervention cohorts; recruitment centre for multi-centre cohorts; socio-economic status and urban/rural residence, as deemed appropriate)
* Model 3: M2 + red and processed meat, fruit and vegetable, potatoes, fish, legume, egg, cereal, whole grain, coffee, tea, sugar- and artificially-sweetened beverages and cooking fats. For analysis by subtype of nuts, model 2 will also be mutually adjusted for each other types of nut.
* Model 4: M3 + body mass index Subgroups analyses will be performed based on age, sex, race, educational level, physical activity level, smoking status, body weight status, hypercholesterolemia and diabetes status at baseline.

All analyses will be restricted to participants with complete data on age, sex, nut consumption, or the disease of interest. The missing data will be handled as follows: a) If there is more than 20% missing data for a covariate, the variable will not be included in the adjustment models; b) If there is 20% or less missing data, for continuous variables, the media should be imputed, and for categorical variables, an additional missing category should be created and used it in the models to avoid losing count or power.

Once all the cohorts have provided the summary statistics, and the results have been verified and harmonized, they will be combined by inverse-variance weighted random effects meta-analyses (DerSimonian and Laird procedure). The between-study variance will be used to assess heterogeneity. To ensure the reliability of the results, additional meta-analyses will be conducted by systematically excluding one cohort at a time. Statistical meta-analyses will be performed using Stata/SE software, version 18.0 (StataCorp, College Station, TX).

ELIGIBILITY:
Inclusion Criteria:

Prospective studies with:

* Dietary data (consumption of nuts, both overall and/or by type) from semiquantitative food frequency questionnaires
* Available data on at least two of the health outcomes of interest
* More than 1,000 adult participants (aged 18 and over)
* A minimum of five years of median follow-up

Exclusion Criteria:

* Prospective studies determining the consumption of nuts in combination with other food groups (e.g., seeds) or with other nut forms (e.g., butter or oil)
* Participants with:
* Missing data on age, sex, and nut consumption.
* Extreme energy intakes (<600 or >3,500 kcal for women and <800 or >4,200 kcal for men)
* The disease of interest at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants from Cohorts larger than 5000 participants and with at least a mean of 5 years of follow-up
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Type-2 diabetes incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
CVD incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Coronary health disesase incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Stroke incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Total cancer incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
All-cause mortality rate | Minimum of five years of median follow-up
  National death registry, self-reported or medication check
CVD-mortality rate, | Minimum of five years of median follow-up
  National death registry, self-reported or medication check
Cancer-mortality rate | Minimum of five years of median follow-up
  National death registry, self-reported or medication check

SECONDARY OUTCOMES:
Total dementia incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Undefined dementia incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Alzheimer's disease incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check
Parkinson's disease incidence | Minimum of five years of median follow-up
  Medical diagnosis, self-reported or medication check

CONTACTS AND LOCATIONS:
Locations (2):
- Department of Public Health, Section of Epidemiology, Copenhagen, Denmark
- Human Nutrition Unit - Alimentació, Nutrició, Desenvolupament i Salut Mental (ANUT-DSM)., Reus, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No
Individual cohorts only send summary data as per the harmonised analysis plan to the study leads. Therefore, the individual participant data remain with the individual cohorts.